CLINICAL TRIAL: NCT03853369
Title: Post-marketing Registration Study of Nifekalant Hydrochloride (NIF) Injection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Peking University First Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: NPMR01/ GUSU18002
Record Dates: First submitted 2019-02-13; First posted 2019-02-25 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-02

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation
Keywords: ventricular tachycardia; ventricular fibrillation
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation | interventions — nifekalant; Injections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Nifekalant hydrochloride — Treatment is not limited. Patients who have used or will use Nifekalant hydrochloride.
  Other Names: Nifekalant Hydrochloride for Injection

SUMMARY:
Retrospective and Prospective single arm, observational study to evaluate efficacy and safety of NIF in the treatment of ventricular tachycardia and ventricular fibrillation. The information registration of the target population will be collected with the hospital HIS system or LIS system.

DETAILED DESCRIPTION:
Subjects enrolled in the retrospective study may be enrolled in a prospective study if the study drug is re-used, but in the end only the most-registered case of the subject would be collected.

The recommended treatment plan for this study is from the usage and dosage of NIF. The clinician can make appropriate adjustments to the specific usage and dosage according to the patient's condition.

Load dose: Adults usually use 0.3mg/kg each time, under continuous ECG monitoring, the injection should be completed within 5 minutes, and the maximum dose should not exceed 0.5 mg/kg.

Maintenance dose: After load injection, the adult routine dose is 0.4 mg/kg/h under continuous ECG monitoring. The dosage could be appropriately increased or decreased according to the patient's reaction, but the maximum dose should not exceed 0.8 mg/kg/h.

ELIGIBILITY:
Inclusion Criteria:

* Patients with life-threatening ventricular tachycardia or ventricular fibrillation in cases where other drugs are ineffective or inoperable.
* Patients who have received or are about to receive Nifekalant Hydrochloride for treatment according to the instructions.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with life-threatening ventricular tachycardia or ventricular fibrillation in cases where other drugs are ineffective or inoperable.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
The rate of termination / prevention of ventricular tachycardia / ventricular fibrillation attack and relapse. | From the beginning of the administration to 48 hours after the end of the administration.
  The efficiency during the treatment and observation periods, including the rate of termination / prevention of ventricular tachycardia / ventricular fibrillation attack and relapse.

SECONDARY OUTCOMES:
Number of Participants with adverse events | From the beginning of the administration to 48 hours after the end of the administration.
  Number of Participants with Tdp, ventricular tachycardia or ventricular fibrillation.
Heart rate | 3 days before the beginning of the administration to 48 hours after the end of the administration.
  The subjects' heart rate will be recorded and the abnormalities will be analyzed.
The survival rate | 30 days after the end of administration.
  The 30 days survival rate.
Blood pressure | 3 days before the beginning of the administration to 48 hours after the end of the administration.
  Both systolic and diastolic pressures will be assessed during the study period.
Respiratory rate | 3 days before the beginning of the administration to 48 hours after the end of the administration.
  The respiratory status of all subjects will be recorded the incidence of abnormalities will be calculated.
Body temperature | 3 days before the beginning of the administration to 48 hours after the end of the administration.
  The subjects' temperatures will be recorded and the abnormalities will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, Principal Investigator — Peking University First Hospital; Jing Zhou, Principal Investigator — Peking University First Hospital; Min Yi Cui, Principal Investigator — Peking University First Hospital; Xin Hu, Principal Investigator — Beijing Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No